CLINICAL TRIAL: NCT04716959
Title: A Randomized Controlled Trial of Prepectoral Versus Subpectoral Prosthetic Breast Reconstruction
Brief Title: Comparing Two Different Surgical Techniques for Breast Reconstruction
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study recommended for closure
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-565
Record Dates: First submitted 2021-01-19; First posted 2021-01-20 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Breast Reconstruction
Keywords: Prosthetic; Breast tissue expander; 20-565

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prepectoral Prosthetic Breast Reconstruction (Experimental)
  Interventions: Procedure: Prepectoral Prosthetic Breast Reconstruction
- Subpectoral Prosthetic Breast Reconstruction (Active Comparator)
  Interventions: Procedure: Subpectoral Prosthetic Breast Reconstruction

INTERVENTIONS:
Procedure: Prepectoral Prosthetic Breast Reconstruction — The prepectoral approach involves placing the tissue expander on top of the pectoralis muscle.
  Arms: Prepectoral Prosthetic Breast Reconstruction
Procedure: Subpectoral Prosthetic Breast Reconstruction — The subpectoral approach involves placing the tissue expander under the pectoralis muscle with or without acellular dermal matrix (ADM).
  Arms: Subpectoral Prosthetic Breast Reconstruction

SUMMARY:
The purpose of this study is to compare two standard techniques for breast reconstruction-the prepectoral technique and the subpectoral technique. Again, the prepectoral technique involves putting a tissue expander on top of the pectoralis muscle, while the subpectoral technique involves putting a tissue expander under the pectoralis muscle.

The standard approach used at MSK is the subpectoral technique. This study will help researchers find out whether the subpectoral approach is better, the same as, or worse than the prepectoral approach. To decide which approach is better, the researchers will look at which technique causes fewer complications after surgery (for example, infection or the need for a second surgery). Researchers are also interested in seeing which approach causes less pain and use of pain medication after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 21-60 years
* Planning to undergo immediate two stage prosthetic breast reconstruction with TE placement as the first stage.
* Planning to undergo unilateral or bilateral mastectomy.
* Planning to undergo nipple- or skin-sparing mastectomy.
* Mastectomy weight less than 800 grams.
* Adequate mastectomy skin perfusion or patients with adequate perfusion but nonviable mastectomy skin that can be excised (≤ 4 cm) at the defect margins with otherwise adequate perfusion.

Exclusion Criteria:

* Receipt of neoadjuvant chemotherapy for locally advanced breast cancer.
* Presence of preoperative axillary lymph node metastasis.
* Presence of intraoperative sentinel node positivity.
* History of radiotherapy.
* Current smoker.
* Planning to undergo direct-to-implant reconstruction.
* BMI >35.
* Prior sternotomy.

Ages: 21 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Breast Reconstruction
Enrollment: 0 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2021-12-13 (Actual)

PRIMARY OUTCOMES:
major perioperative complications | 90 days
  90-day major complications for tissue expanders (i.e., infection, explantation, and reoperation for mastectomy flap necrosis):
  * Infection: any event requiring restart of antibiotics (oral or intravenous) following completion of initial perioperative antibiotics or an admission to the hospital for cellulitis.
  * Explantation: need for tissue expander removal for any cause.
  * Reoperation: skin excision performed in either the clinic or the main operating room for mastectomy skin flap necrosis.

SECONDARY OUTCOMES:
minor complications | 90 days
  Minor complication for tissue expanders is defined as: Seroma: clinically significant non-infected fluid collection requiring either needle aspiration or drain replacement

CONTACTS AND LOCATIONS:
Overall Officials: Evan Matros, MD, MMSc, MPH, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering BaskingRidge (Consent and Followup), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent and Followup), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent and Followup ), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Consent and Followup), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent and Followup), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Consent and Followup), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm